CLINICAL TRIAL: NCT04741555
Title: The Effect of Preoperative Neutrophil / Lymphocyte Ratio and Uric Acid Values on Short and Long Term Mortality in Patients Undergoing Open Heart Surgery
Brief Title: The Effect of Preoperative Values on Mortality in Patients Undergoing Open Heart Surgery
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ali AKDOĞAN, assistant professor, Karadeniz Technical University
Other Study IDs: 2020/295
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Mechanical Ventilation; Coronary Bypass Surgery; Postoperative Complications
Keywords: neutrophil / lymphocyte ratios; uric acid level; mortality; coronary bypass surgery; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Open heart surgeries are one of the major and complicated surgeries performed frequently in the world due to the prolongation of life expectancy and developments in medicine. As a result of these operations, not only the heart and vessels, but also all organs and systems depending on the systemic circulation are affected. Some biological inflammation markers have been determinant in determining cardiovascular risk. High neutrophil count was associated with increased mortality, while low lymphocyte count was a strong constant predictor of mortality. In addition, increased serum uric acid (UA) levels have been found to be associated with obesity, dyslipidemia, and hypertension, which is associated with cardiovascular disease risk. The aim of this study is to investigate the effects of patients who underwent coronary bypass surgery under elective conditions in Karadeniz Technical University Faculty of Medicine between 2008-2020 on in-hospital and 1-year mortality based on preoperative neutrophil / lymphocyte ratios and uric acid values.

DETAILED DESCRIPTION:
Open heart surgeries are one of the major and complicated surgeries performed frequently in the world due to the prolongation of life expectancy and developments in medicine. Mortality rates are decreasing day by day, although more and more additional diseases are present and older patients are taken in open heart surgery. The aim of these surgeries is to reduce the risk of death by correcting existing cardiac pathologies and increasing the quality of life of patients. For this reason, some studies have developed cardiac risk scoring methods in preoperative evaluation in order to predict mortality before surgery, and created a risky group such as advanced age, female gender, decreased left ventricular functions, those who use postoperative intraaortic balloon pumps, and those who receive inotrope support.

Some biological inflammation markers have been determinant in determining cardiovascular risk. High neutrophil count was associated with increased mortality, while low lymphocyte count was a strong constant predictor of mortality. Cardiovascular bypass itself is related to neutrophil activation, highlighting the effects of its high preoperative levels. Increased neutrophil counts are related to blood viscosity and hypercoagulability. Also, decreased lymphocyte count indicates increased physiological stress.

The importance of serum uric acid levels has been stated in many epidemiological studies as a risk factor for cardiovascular diseases. Increased serum uric acid (UA) levels are associated with obesity, dyslipidemia, and hypertension, which is associated with a risk of cardiovascular disease. In another study, it was shown that the risk of cardiovascular mortality and increased serum UA levels were independently and significantly related.

The aim of this study was to examine the short-term (first 30 days) and long-term (1 year) mortality of patients who underwent elective coronary bypass surgery between 2008 and 2020 at the Karadeniz Technical University Faculty of Medicine, based on preoperative neutrophil / lymphocyte ratios and uric acid values. effects will be investigated

ELIGIBILITY:
Inclusion Criteria:

* Elective patients undergoing open heart surgery

Exclusion Criteria:

* Immunodeficiency
* Emergency operations
* Patients whose records could not be accessed and who were excluded from the study group procedure in which they were included for any reason will not be included in the study.
* Patients under 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study was planned as a retrospective (retrospective) study involving patients who underwent elective open heart surgery between January 1, 2008 and December 31, 2020
Sampling Method: Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
neutrophil / lymphocyte ratios | postoperative 2 week
  The effect on postoperative complications of preoperative neutrophil lymphocyte ratio in open heart surgery
neutrophil / lymphocyte ratios | postoperative 1 year
  The effect on mortality of preoperative neutrophil lymphocyte ratio in open heart surgery
uric acid values | postoperative 1 year
  The effect on mortality of preoperative uric acid values in open heart surgery
uric acid values | postoperative 2 week
  The effect on postoperative complications of preoperative uric acid values in open heart surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)